CLINICAL TRIAL: NCT00004893
Title: Evaluation of Novel Therapeutic Agents Against Breast Cancer: An Innovative Randomized Phase II Trial Design
Brief Title: Interleukin-12 in Treating Patients With Metastatic or Recurrent Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-49806; U10CA031946 (NIH); CLB-49806; CDR0000067570 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-03-07; First posted 2004-05-03 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Interleukin-12 Subunit p35

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IL12 Therapy (Experimental): Patients begin therapy no sooner than 3 weeks and no later than 6 weeks since last chemotherapy dose. Patients receive interleukin-12 subcutaneously twice a week. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed at least every 3 months for 1 year. If no progression after 1 year, may be followed as needed for new signs or symptoms and survival for 5 years.
  Interventions: Biological: recombinant interleukin-12
- Observation (No Intervention): Patients are observed for 6 months. If disease progresses during first 6 months, patients may receive interleukin-12 as in arm I. Patients without disease progression within first 6 months may also then receive interleukin-12 as in arm I. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed for toxicity only until interleukin-12 is discontinued.

INTERVENTIONS:
Biological: recombinant interleukin-12
  Arms: IL12 Therapy

SUMMARY:
RATIONALE: Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill breast cancer cells.

PURPOSE: Randomized phase II trial to study the effectiveness of interleukin-12 in treating patients who have metastatic or recurrent breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the activity of interleukin-12 as defined by the percentage of patients who have not progressed after 6 months of therapy. II. Compare percentage of patients who have not progressed after six months with or without treatment regimen. III. Determine time to progression and overall survival in this patient population after this treatment.

OUTLINE: This is a randomized study. Patients are stratified according to disease free interval from primary diagnosis to first metastases (less than 3 years vs 3 years and longer), estrogen receptor status (positive vs negative), and disease status (complete response, partial response, detectable disease, or stable disease). Patients are randomized to one of two treatment arms. Arm I: Patients begin therapy no sooner than 3 weeks and no later than 6 weeks since last chemotherapy dose. Patients receive interleukin-12 subcutaneously twice a week. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed at least every 3 months for 1 year. If no progression after 1 year, may be followed as needed for new signs or symptoms and survival for 5 years. Arm II: Patients are observed for 6 months. If disease progresses during first 6 months, patients may receive interleukin-12 as in arm I. Patients without disease progression within first 6 months may also then receive interleukin-12 as in arm I. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed for toxicity only until interleukin-12 is discontinued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic or recurrent breast cancer (not confined to breast) One prior induction chemotherapy regimen for recurrent or metastatic disease (4 weeks of treatment for 4-6 courses) resulting in stable disease, partial response, or complete response Pleural or peritoneal effusion palliated by induction chemotherapy allowed No uncontrolled brain metastases Previously treated brain metastases allowed if: No evidence of progression for at least 3 months following radiotherapy and/or surgical treatment AND At least 30 days since dexamethasone or other corticosteroids AND Other metastatic site exists No bone marrow or brain as only sites of metastases No meningeal disease Hormone receptor status Estrogen receptor status known

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Menopausal status: Not specified Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Hemoglobin at least 9 g/dL (transfusion or epoetin alfa allowed) Platelet count at least 100,000/mm3 Hepatic: SGOT/SGPT no greater than 1.5 times upper limit of normal (ULN) Albumin at least 3.0 g/dL Bilirubin no greater than 1.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Creatinine clearance at least 60 mL/min Other: No other active malignancy except nonmelanoma skin cancer Not pregnant or nursing Fertile patients must use effective contraception No inflammatory bowel disease or active gastric ulcer No prior autoimmune disease or immunodeficiency syndrome

PRIOR CONCURRENT THERAPY: Biologic therapy: See Chemotherapy No concurrent interleukin-11 Chemotherapy: See Disease Characteristics No concurrent chemotherapy Prior chemotherapy with bone marrow progenitor support (bone marrow transplant and/or peripheral blood stem cell support) allowed in adjuvant setting only (not for metastases) Endocrine therapy: Prior hormone therapy for breast cancer allowed No concurrent hormones allowed except for non-cancer or cancer treatment related conditions (e.g. insulin for diabetes) No concurrent dexamethasone or other steroidal antiemetics Radiotherapy: Prior radiotherapy allowed No concurrent radiotherapy Surgery: Not specified Other: Prior bisphosphonate therapy allowed if started at least 3 months before study No initiation of bisphosphonate therapy during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1999-12; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
disease progression | at 6 months

SECONDARY OUTCOMES:
time to progression | Up to 1 year
overall survival | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F. Hayes, MD, Study Chair — University of Michigan Rogel Cancer Center
Locations (49):
- United States (49):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia